CLINICAL TRIAL: NCT03572608
Title: Clinical Effectiveness of Acupuncture to Increase Pregnancy Success Rates for Women Undergoing in Vitro Fertilization: A Randomized Controlled Trial
Brief Title: Pregnancy Success Rates of Acupuncture for in Vitro Fertilization
Acronym: Acupuncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Yasemin Cayir, Assoc. Prof. Yasemin Cayir, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/120
Record Dates: First submitted 2018-05-28; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Infertility, Female
Keywords: acupuncture; infertility; pregnancy
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Treatment (Experimental): Acupuncture group will receive 3 acupuncture sessions. The first session will be one week before embryo transfer. The second session will be 30 minute before embryo transfer. And the last session will be 30 minute after embryo transfer.
  Interventions: Other: Acupuncture treatment
- Control Group (No Intervention): Control Group will not receive any acupuncture session before or after embryo transfer.

INTERVENTIONS:
Other: Acupuncture treatment — Classical acupuncture points will be used without a formal traditional Chinese medicine diagnosis in the intervention group. Neither manual needle stimulation nor moxibustion will used. The needles will left in place for 30 min and de qi was not sought. The points will be selected bilateral Heart-7, bilateral Large Intestine-4, Governing Vessel-20 and ear shenmen for the first session. Bilateral Conception Vessel-3,4,6, bilateral Liver-3, bilateral Stomach-30, bilateral Spleen-6, bilateral Governing Vessel-20 will be used for the second session. Bilateral Large Intestine-4, bilateral Spleen-6,9, bilateral Stomach-36 will be used for the last session. All acupuncture points will be selected and localized on the basis of the WHO Standardised Acupuncture Point Location.
  Arms: Acupuncture Treatment

SUMMARY:
This study evaluates the effectiveness of acupuncture on pregnancy success before embryo transfer in IVF treatment in female infertile patients. Half of participants will receive acupuncture sessions before embryo transfer, while the other half will not receive.

DETAILED DESCRIPTION:
Acupuncture is used for many health problem all around the World. WHO reported that acupuncture can have benefit in female infertility treatment. However, there is no enough evidence about effectiveness of acupuncture treatment in the infertility.

ELIGIBILITY:
Inclusion Criteria:

* To have unexplained infertility
* To go in vitro fertilization treatment
* To give permission by informed consent form

Exclusion Criteria:

* Below age of 18 and above age of 45
* To have secondary infertility
* To reject completing informed consent form

Ages: 23 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation
Enrollment: 120 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
pregnancy | 2 weeks after the treatment
  positive betaHCG

SECONDARY OUTCOMES:
Anxiety level | Through study completion, 2 weeks after the protocol
  STAI-1 Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Bunyamin Borekci, Study Chair — Ataturk University
Locations (1):
- Ataturk University Hospital, Erzurum, Turkey (Türkiye)